CLINICAL TRIAL: NCT02405104
Title: Analgetic Effects of Chlorzoxazone in Total Hip and Knee Arthroplasty
Brief Title: Chlorzoxazone in Hip and Knee Arthroplasty
Acronym: chlorzoxazon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Principal Investigator, Mogens Laursen, MD PhD, Associate Professor, PhD, Northern Orthopaedic Division, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ON-151-MU-Klorz
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis of Hip; Osteoarthritis, Knee
Keywords: osteoarthritis; hip; knee; total hip arthroplasty; total knee arthroplasty; post operative pain management
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis | interventions — Chlorzoxazone; Tacrine; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- THA+Klorz (Active Comparator): All patients in this arm are treated surgically with a THA and medically with Chlorzoxazone
  Interventions: Drug: chlorzoxazone; Procedure: THA
- THA+Placebo (Placebo Comparator): All patients in this arm are treated surgically with a THA and medically with placebo
  Interventions: Drug: Placebo; Procedure: THA
- TKA+Klorz (Active Comparator): All patients in this arm are treated surgically with a TKA and medically with Chlorzoxazone
  Interventions: Drug: chlorzoxazone; Procedure: TKA
- TKA+Placebo (Placebo Comparator): All patients in this arm are treated surgically with a TKA and medically with placebo
  Interventions: Drug: Placebo; Procedure: TKA

INTERVENTIONS:
Drug: chlorzoxazone — ATC-code: M03BB03
  Other Names: ATC-code M03BB03
  Arms: THA+Klorz; TKA+Klorz
Drug: Placebo — Placebo
  Arms: THA+Placebo; TKA+Placebo
Procedure: THA — Surgical treatment of osteoarthrosis in the hip, by replacement.
  Other Names: Total Hip Arthroplasty
  Arms: THA+Klorz; THA+Placebo
Procedure: TKA — Surgical treatment of osteoarthrosis in the knee, by replacement.
  Other Names: Total Knee Arthroplasty
  Arms: TKA+Klorz; TKA+Placebo

SUMMARY:
The purpose of this study is to elucidate whether patients operated with THA and TKA can benefit from treatment with chlorzoxazone.

DETAILED DESCRIPTION:
Introduction and rationale Background Modern treatment of pain following surgery based on multimodal analgesic strategy where the pain system different points of attack struck with different types analgesics. This also tries to reduce the consumption of opioids associated with frequent side effects like nausea, vomiting, constipation, difficulty urinating, weather stretch problems and Lethargy.

But in spite of intense research over the last decades, is pain after arthroplastic surgery in hip (total hip arthroplasty (THA)) or knee (total knee replacement (TKA)) continue a significant clinical problem. It is a current clinical assumption that patients with pain in the hip or knee region immediately after TKA or THA have tense muscles, which reinforces pain behavior. The mechanism for such muscle tension is not fully understood.

For many years the investigators have been on Danish orthopedic departments dealt with these patients with postoperative pain after major joint prosthesis operations with the muscle relaxant chlorzoxazone. On some sections included in the standard chlorzoxazone prescriptions for pain after hip and knee replacement.

chlorzoxazone has for many years been marketed for the treatment of pain in skeletal muscle by inhibition of mono- and polysynaptic reflexes in the CNS. The muscle relaxing effect is mediated by inhibitory effects on spinal polysynaptic reflexes. In placebo-designed clinical studies of chlorzoxazone's beneficial effect on heterogeneous groups of patients with spasticity, motor neuron syndromes, as well as muscle pain and spasm of peripheral musculoskeletal diseases have not been able to demonstrate no significant analgesic effect; chlorzoxazone have also failed to show pain-relieving effect in the treatment of back pain It is remarkable that in spite of the widespread use of chlorzoxazone not can be found only one study of chlorzoxazone used as adjuvant pain relieving treatment after hip or knee surgery (or other orthopaedic treatment). The current clinical practice is therefore made on purely empirical basis. The effect must be considered as uncertain, but may in some cases be indicated, most often as an adjunct to other therapy, for example analgesics, anti-inflammatory agents, physiotherapy or even training. In such cases, regarded chlorzoxazone be an alternative to benzodiazepines. There is therefore a need for a prospective, randomized, double-blind, placebo-controlled study evaluating the potential analgesic effect of chlorzoxazone. In this intervention study is the selected dosage of chlorzoxazone set at based on the recommendation of the Danish Medicines Information A / S 7 (http://pro.medicin.dk/Medicine / Preparations / 638) and Takeda Pharma A / S. The latter produces chlorzoxazone. The recommendation is based on our current knowledge of chlorzoxazones pharmacodynamic and pharmacokinetic properties. chlorzoxazone given in this study as tablet chlorzoxazone, 250 mg, 3 times daily for the first seven postoperative days. Adverse reactions to chlorzoxazone are well known. They are relatively few, mostly mild and transient. The most frequent adverse events related to chlorzoxazone, fatigue and dizziness (about 1-10% of patients) Adverse reactions are to some extent overlapping with the side effects that are related to the perioperative opioid treatment. It is therefore possible that the frequency of adverse events overall is reduced if chlorzoxazone found to be analgesic (and opioid-sparing). Patients will be hospitalized for a minimum of two nights after surgery and thus be close observation in the period in which the risk of side effects is greatest. At the same time, all patients undergo standardized adverse event registration. If, contrary to expectations unexpected or unacceptable side effects medication will promptly be interrupted. The study involves a group of patients (THA and TKA), which is an important clinical pain problem. All of these patients receive a well-implemented and evidence-based treatment. Thus, anesthesia, analgesia and surgical procedure standardized for all patients receiving concomitant consequences usual principles of early mobilization 8; 9th The planned randomized, double-blind, placebo-controlled design in which all patients receive the same and standardized interventions, enabling the best possible evaluation of modality under study intervention with chlorzoxazone vs. placebo). The level of pain after surgery as the primary endpoint, recorded by means of a well-tested and validated tool (visual analog scale (VAS)) 48 hours after operation. The current study could contribute to a clarification of the postoperative analgesic effect of chlorzoxazone immediately after THA and TKA. As secondary endpoints, the patients functional level be determined Oxford Hip / Knee Score 7 days after surgery. Furthermore, a number of tertiary parameters related to pain, function and side effect profile be determined as shown in Table 1. Evidence in this area will be of immediate benefit to patients operated with THA and TKA - and maybe for other surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Planned primary unilateral THA or TKA
* Patients (male/female) ≥ 18 år
* Patients giving written informed consent and authority.
* Patients receiving spinal anaesthesia

Exclusion Criteria:

* Patients with intolerance to trial medications
* Rejection of or contraindicated spinal anaesthesia
* Patients with rheumatoid arthritis.
* Patients with Body Mass Index (BMI) ≥ 35
* Patients that do not read or write Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Pain after 5 meter walk | 24 hours post OP
  VAS-score

SECONDARY OUTCOMES:
Oxford Hip/Knee score | 7 days post OP
  standardized functional and pain score
Pain at rest | until 12 months after surgery
  VAS
worst pain for the last 24 hours | until 12 months after surgery
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Mogens Laursen, MD, PhD, Principal Investigator — Northern Orthopaedic Division, Denmark
Locations (1):
- Northern Orthopaedic Division, Clinic Farsø, Aalborg University Hospital, Farsø, Northern Jutland, Denmark